CLINICAL TRIAL: NCT07035587
Title: Diagnosis of Multiple Cancer and Monitoring of Minimal Residual Tumors After Treatment Using Blood and High-Sensitivity Genetic Analysis Techniques
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2024-0702
Record Dates: First submitted 2025-06-15; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Lung Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Ovarian Neoplasms; Stomach Neoplasms; Neoplasm Micrometastasis; Neoplasms
MeSH Terms: conditions — Lung Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Ovarian Neoplasms; Stomach Neoplasms; Neoplasm Micrometastasis; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer Patient Group: Patients diagnosed with stage I-IV pancreatic, lung, colorectal, ovarian, esophageal, gastric, hematologic, breast, renal, bladder, or prostate cancer, including those undergoing surgery or chemotherapy. Blood samples will be collected serially before and after treatment and during outpatient follow-up visits. Samples will be analyzed for circulating tumor DNA (ctDNA), cell-free DNA (cfDNA), RNA, and protein profiles to monitor tumor dynamics and evaluate diagnostic accuracy. Tissue biopsies will be used to compare tumor-specific mutations with those detected in ctDNA.
  Interventions: Other: Serial Blood Sampling for Molecular Profiling
- Control Group: Healthy individuals or patients with asymptomatic gallstones or benign colon polyps, or those undergoing routine health screening without a history of cancer. A single blood sample will be collected for cfDNA, RNA, and protein analysis. These samples will serve as comparators to assess molecular differences between non-cancer and cancer populations.
  Interventions: Other: One-Time Blood Sampling for Molecular Profiling

INTERVENTIONS:
Other: Serial Blood Sampling for Molecular Profiling — Cancer patients will undergo serial peripheral blood sampling at baseline (prior to surgery or chemotherapy), after treatment, and during follow-up visits. Blood samples will be analyzed for circulating tumor DNA (ctDNA), cell-free DNA (cfDNA), RNA, and protein biomarkers. The purpose is to detect variant allele frequency (VAF) and evaluate its relationship with tumor dynamics and treatment outcomes, including recurrence and survival.
  Groups: Cancer Patient Group
Other: One-Time Blood Sampling for Molecular Profiling — Control participants, including individuals with asymptomatic gallstones, benign polyps, or those undergoing health screening, will provide a one-time peripheral blood sample. The sample will be analyzed for cfDNA, RNA, and protein biomarkers and used as a baseline reference to compare molecular characteristics between non-cancer and cancer groups.
  Groups: Control Group

SUMMARY:
This is a combined prospective and retrospective observational study aiming to validate a highly sensitive and specific blood-based method for the early diagnosis and post-treatment monitoring of multiple cancers. The study leverages a newly developed sequencing method to improve the detection of circulating tumor DNA (ctDNA) in blood, focusing on enhancing sensitivity and specificity in clinical applications.

The study targets patients with ovarian, lung, pancreatic, colorectal, esophageal, breast, kidney, bladder, and gastric cancer, as well as healthy controls with asymptomatic gallstones, benign polyps, or individuals undergoing routine medical screening. Blood samples will be analyzed for cell-free DNA (cfDNA), RNA, and protein profiles. A key objective is to determine how much the newly developed method increases the sensitivity and specificity of ctDNA detection, especially in early-stage cancers and minimal residual disease (MRD) after treatment.

The method evaluates the variant allele frequency (VAF) of ctDNA to detect residual disease and track tumor dynamics. Serial blood sampling will be conducted before and after surgery or chemotherapy and during follow-up outpatient visits in cancer patients, while one-time sampling will be done for controls. Additionally, tissue biopsies collected during surgery will be used to analyze concordance between tumor-specific mutations and those found in ctDNA.

Primary outcome measures include quantitative differences in ctDNA or RNA levels between cancer and control groups. Secondary outcomes assess the clinical correlation between changes in ctDNA VAF and patient outcomes such as recurrence and survival. Statistical tools including ROC curve analysis, Cox regression, and log-rank tests will be used to quantify performance.

This study seeks to establish a clinically robust, non-invasive diagnostic tool that enables earlier detection and more precise treatment decisions, while potentially reducing physical, psychological, and socioeconomic burdens related to cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years
* Voluntarily agreed to participate and provided informed consent
* Able to donate blood without health risks
* Underwent or is scheduled to undergo surgery or chemotherapy for therapeutic purposes for cancer (for cancer group)
* Diagnosed with one of the following cancers: ovarian, lung, pancreatic, colorectal, esophageal, breast, bladder, kidney, or gastric cancer
* Control group: asymptomatic individuals with gallstones or benign polyps, or subjects undergoing routine health screenings
* Control group must have confirmed benign findings through imaging (ultrasound, CT, LDCT, colonoscopy)

Exclusion Criteria:

* Age < 19 years
* Patients with mental retardation or severe psychiatric disorders affecting informed consent
* History of HIV, HTLV, or syphilis infection
* History of other malignancy within 5 years (for cancer group)
* No somatic mutation detected in tumor or pre-treatment cfDNA (for cancer group)
* Control group with any past or current cancer diagnosis
* Control group with high-grade adenoma, symptomatic gallstones/polyps, or recent (<6 months) abdominal surgery
* Pregnant or breastfeeding women
* Any other reason deemed inappropriate by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from patients and screening subjects at Yonsei University Health System (Severance Hospital, Yonsei Cancer Center, and affiliated check-up centers in Seoul, South Korea). The study population includes individuals diagnosed with ovarian, lung, pancreatic, colorectal, esophageal, breast, bladder, kidney, or gastric cancers, either newly diagnosed or post-treatment. The control group includes individuals with asymptomatic gallstones, benign polyps, or those undergoing routine health screenings. All participants must be 19 years or older and able to provide informed consent for blood collection and data/sample usage.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2029-07-28 (Estimated); Study Completion 2029-07-28 (Estimated)

PRIMARY OUTCOMES:
Difference in significantly detected ctDNA Variant Allele Frequency (VAF) between Cancer Patients and Controls | At baseline and up to 66 months post-enrollment
  Quantitative measurement of significantly detected ctDNA variant allele frequency (VAF) in plasma samples from blood collected at baseline and follow-up visits (every 3-12 months up to 2 years) will be used to assess sensitivity and specificity of the developed sequencing method in detecting cancer-associated mutations. ROC curve analysis will be applied to determine the method's diagnostic performance (e.g., AUC).

SECONDARY OUTCOMES:
Correlation between ctDNA VAF and Clinical Outcomes (Recurrence and Survival) | Baseline and follow-up at 3-12 month intervals, up to 36 months
  To evaluate the relationship between ctDNA variant allele frequency (VAF) changes and patient clinical outcomes, including recurrence free and overall survival. Longitudinal VAF trends will be correlated with disease progression. Additionally, concordance between ctDNA mutations and matched tumor tissue mutations will be assessed. In patients receiving chemotherapy, detection of resistance-related mutations in ctDNA will be evaluated for associations with treatment outcomes. Survival analysis will use Cox regression and log-rank tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pharmacology, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol